CLINICAL TRIAL: NCT00557960
Title: A Phase IIIb Study to Evaluate the Efficacy and Time Course of Treatment With ADDERALL XR and STRATTERA Compared to Placebo on Simulated Driving Safety and Performance and Cognitive Functioning in Adults With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: ADDERALL XR (Mixed Salts of a Single-entity Amphetamine) and STRATTERA ( Atomoxetine Hydrochloride) Compared to Placebo on Simulated Driving Safety and Performance and Cognitive Functioning in Adults With ADHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SLI381-316
Record Dates: First submitted 2007-11-09; First posted 2007-11-14 (Estimated); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — SLI381; Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Mixed salts of a single-entity amphetamine
  Other Names: ADDERALL XR
Drug: Atomoxetine hydrochloride
  Other Names: STRATTERA

SUMMARY:
Evaluate the efficacy of treatment with ADDERALL XR and STRATTERA compared to placebo on simulated driving safety and performance of young adults with ADHD as measured by Driving Safety Scores derived by the Driving Simulator.

ELIGIBILITY:
Inclusion Criteria:

* primary diagnosis of ADHD
* not naive to pharmacologic ADHD treatment
* valid driver's license with a minimum of 3 years driving experience

Exclusion Criteria:

* recent history of drug dependence or substance use disorder
* any specific cardiac condition that would, in the opinion of the investigator, require exclusion
* history of seizure in last 2 years, tic disorder or Tourette's disorder
* female subject is pregnant or lactating

Ages: 19 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2004-02-25 (Actual); Primary Completion 2004-10-25 (Actual); Study Completion 2004-10-25 (Actual)

PRIMARY OUTCOMES:
Overall Driving Safety Score derived by the driving simulator | Weeks 3 & 6

SECONDARY OUTCOMES:
Driving Safety Scores at individual time points | 2, 7, and 12 hours post-dose at Weeks 3 & 6
Cog-Screen Aviator Predictor Score, ADHD-RS, CGI, Self-rating of driving simulator performance questionnaire | Weeks 3 & 6
AEs, laboratory screens, PE, vital signs, ECG | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Washington Neuropsychological Institute, LLC, Washington D.C., District of Columbia, United States

REFERENCES:
- [Result] Kay GG, Michaels MA, Pakull B. Simulated driving changes in young adults with ADHD receiving mixed amphetamine salts extended release and atomoxetine. J Atten Disord. 2009 Jan;12(4):316-29. doi: 10.1177/1087054708322986. Epub 2008 Sep 24. PMID 18815438
- See also: FDA Recall Information — http://www.fda.gov/opacom/7alerts.html